CLINICAL TRIAL: NCT03915756
Title: Postoperative Drainage in Total Knee Arthroplasty in the Presence of Tranexamic Acid: a Clinical Trial
Brief Title: Postoperative Drainage in Total Knee Arthroplasty in the Presence of Tranexamic Acid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Beatriz Ângelo (Other)
Responsible Party: Principal Investigator, Afonso Cardoso, Principal Investigator, Hospital Beatriz Ângelo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0389
Record Dates: First submitted 2019-04-12; First posted 2019-04-16 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee replacement; Blood loss; Wound drainage
MeSH Terms: conditions — Osteoarthritis, Knee; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With drain (Experimental): Participants who received a drain during surgery
  Interventions: Procedure: Drainage of surgical wound
- Without drain (No Intervention): Participants who did not receive a drain during surgery

INTERVENTIONS:
Procedure: Drainage of surgical wound — Introduction of a drain before full fascial closure
  Arms: With drain

SUMMARY:
The investigator's aim with this study is to address, with the new paradigm of tranexamic acid, the role of wound drainage following total knee arthroplasty in blood loss, blood transfusion requirements and functional recovery

DETAILED DESCRIPTION:
All participants will attend a preoperatory appointment with an anaesthesiologist where preoperative haemoglobin will be optimized (Hg > 13 g/L).

Randomization will be done by opening a closed envelop with the selected group from a bag at the time of wound closure.

Collected preoperative information will include age, gender, weight, height, body-mass index, underlying diseases, operated side, haematocrit, haemoglobin level, midpatellar knee circumference and range of movement. Blood work was performed within 1 hour of the beginning of the surgery. Clinical parameters will be collected before anaesthesia.

In all cases, the surgeon will perform a medial parapatellar approach with a standard incision with the participants in the supine position. The SIGMA PFC total knee system (DePuy, Warsaw, In) and its posterior-stabilized design with a rotatory platform will be used. All participants will be under a subarachnoid spinal block.

A tourniquet will be used (pressure of 350 mmHg) from the beginning of the surgery and deflated for haemostasis before wound closure. At this time, before complete water-tight fascial closure, the patients will be allocated to group With or Without drain as described, and a drain will be placed in a subfascial position. The drain will be left clamped for 1 hour and will be left in place for 24 hours. Compressive dressings will be applied at the end of the surgery. Continuous passive motion will be started within 24 hours of surgery (0-60°, progressing as tolerated).

In all participants, about 30min before tourniquet release, intravenous tranexamic acid will be used with an initial bolus of 10 mg/kg administered in 10min followed by a perfusion of 10mg/kg over 4h. For postoperative analgesia, a femoral triangle and a popliteal block (anterior approach) will be done in all participants.

A standard fluid therapy of a balanced crystalloid solution (perfusion 10ml/kg/h) will be administered to all patients. After tourniquet release, during haemostasis and in the recovery room, an eventual need of increasing fluid therapy perfusion or a bolus will be noted in the patient's file.

Hidden blood loss will be calculated according to the haemoglobin balance method as it suggested to be the most reliable method. Total blood volume will be calculated as described by Nadler et al.

The normality of the data will be tested with the Shapiro-Wilk test/Kolmogorov-Smirnov test. The data will be compared and analyzed using Student's t-test for independent samples, or the Mann-Whitney test, according to the normality of the data. The correlation of data will be analyzed with the Pearson or Spearman correlation coefficient according to its normality. Nominal variables will be compared using the chi-square test. P-values less than 0.05 will be considered significant. Dedicated statistical software (SPSS version 21, SPSS Inc., Chicago, USA) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients admitted to perform a primary unilateral total knee arthroplasty

Exclusion Criteria:

* Contraindication to take tranexamic acid
* hematologic disease with a higher risk of bleeding
* abnormal coagulation tests
* refusal of blood transfusions
* inadequate preoperatory optimization
* deformity >15⁰ of varus or valgus

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Total RBC loss | 96 hours
  Total red blood cells loss after surgery
Total RBC loss | 24 hours
  Total red blood cells loss after surgery
Total RBC loss | 1 hour
  Total red blood cells loss after surgery
Blood transfusion requirements | 96 hours
  Blood transfusions requirements
Knee Society Score score | 14 days
  Knee Society Score measuring function of Knee (0-100 total score, higher values, better outcome)

SECONDARY OUTCOMES:
Haematocrit level | 1 hour
  Haematocrit level
Haematocrit level | 24 hours
  Haematocrit level
Haematocrit level | 96 hours
  Haematocrit level
Haemoglobin level | 1 hour
  Haemoglobin level
Haemoglobin level | 24 hours
  Haemoglobin level
Haemoglobin level | 96 hours
  Haemoglobin level
Surgery duration | 0hour
  Surgery duration (min)
Length of skin incision | 0 hour
  Length of skin incision
Tourniquet duration | 0 hour
  Tourniquet duration (min)
Surgical blood loss | 0 hour
  Surgical blood loss (mL)
Iron | 96 hours
  Iron products used
Transfusion reactions | 96 hours
  Transfusion reactions
Drain volume | 24 hours
  Drain volume (mL)
MKC | 48 hours
  Midpatellar Knee Circumference (cm)
MKC | 96 hours
  Midpatellar Knee Circumference (cm)
MKC | 14 days
  Midpatellar Knee Circumference (cm)
ROM | 48 hours
  Range of motion (°)
ROM | 96 hours
  Range of motion (°)
ROM | 14 days
  Range of motion (°)
Fluidotherapy excess | 96 hours
  Fluidotherapy excess (mL)
Wound complications (i. e., wound dehiscence, infection) | 14 days
  Wound complications (i. e., wound dehiscence, infection)
Lower leg deep vein thrombosis | 14 days
  Lower leg deep vein thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Afonso Cardoso, Principal Investigator — Hospital Beatriz Angelo
Locations (1):
- Hospital Beatriz Angelo, Loures, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] NIH Consensus Panel. NIH Consensus Statement on total knee replacement December 8-10, 2003. J Bone Joint Surg Am. 2004 Jun;86(6):1328-35. doi: 10.2106/00004623-200406000-00031. No abstract available. PMID 15173310
- [Background] Banerjee S, Kapadia BH, Issa K, McElroy MJ, Khanuja HS, Harwin SF, Mont MA. Postoperative blood loss prevention in total knee arthroplasty. J Knee Surg. 2013 Dec;26(6):395-400. doi: 10.1055/s-0033-1357491. Epub 2013 Oct 11. PMID 24122437
- [Background] Huang GP, Jia XF, Xiang Z, Ji Y, Wu GY, Tang Y, Li J, Zhang J. Tranexamic Acid Reduces Hidden Blood Loss in Patients Undergoing Total Knee Arthroplasty: A Comparative Study and Meta-Analysis. Med Sci Monit. 2016 Mar 10;22:797-802. doi: 10.12659/msm.895571. PMID 26961597
- [Background] Wang H, Shen B, Zeng Y. Comparison of topical versus intravenous tranexamic acid in primary total knee arthroplasty: a meta-analysis of randomized controlled and prospective cohort trials. Knee. 2014 Dec;21(6):987-93. doi: 10.1016/j.knee.2014.09.010. Epub 2014 Oct 23. PMID 25450009
- [Background] Zhang Y, Zhang JW, Wang BH. Efficacy of tranexamic acid plus drain-clamping to reduce blood loss in total knee arthroplasty: A meta-analysis. Medicine (Baltimore). 2017 Jun;96(26):e7363. doi: 10.1097/MD.0000000000007363. PMID 28658157
- [Background] Liao L, Chen Y, Tang Q, Chen YY, Wang WC. Tranexamic acid plus drain-clamping can reduce blood loss in total knee arthroplasty: A systematic review and meta-analysis. Int J Surg. 2018 Apr;52:334-341. doi: 10.1016/j.ijsu.2018.01.040. Epub 2018 Feb 3. PMID 29408472
- [Background] Craik JD, Ei Shafie SA, Kidd AG, Twyman RS. Can local administration of tranexamic acid during total knee arthroplasty reduce blood loss and transfusion requirements in the absence of surgical drains? Eur J Orthop Surg Traumatol. 2014 Apr;24(3):379-84. doi: 10.1007/s00590-013-1206-1. Epub 2013 Mar 14. PMID 23494778
- [Background] Yang Y, Lv YM, Ding PJ, Li J, Ying-Ze Z. The reduction in blood loss with intra-articular injection of tranexamic acid in unilateral total knee arthroplasty without operative drains: a randomized controlled trial. Eur J Orthop Surg Traumatol. 2015 Jan;25(1):135-9. doi: 10.1007/s00590-014-1461-9. Epub 2014 May 10. PMID 24816760
- [Background] Gao FQ, Li ZJ, Zhang K, Sun W, Zhang H. Four Methods for Calculating Blood-loss after Total Knee Arthroplasty. Chin Med J (Engl). 2015 Nov 5;128(21):2856-60. doi: 10.4103/0366-6999.168041. PMID 26521781
- [Background] Nadler SB, Hidalgo JH, Bloch T. Prediction of blood volume in normal human adults. Surgery. 1962 Feb;51(2):224-32. No abstract available. PMID 21936146